CLINICAL TRIAL: NCT03365960
Title: Bioavailability and Pharmacokinetic Parameters of Watermelon (Rind, Flesh and Seeds) Polyphenols in Human Plasma: A Pilot Study to Investigate Relationship to Endothelial Function.
Brief Title: Bioavailability and Pharmacokinetic Parameters of Watermelon (Rind, Flesh and Seeds) Polyphenols
Acronym: WM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: IRB2017-078
Record Dates: First submitted 2017-11-27; First posted 2017-12-08 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Healthy Subjects
Keywords: Watermelon; Watermelon phytochemicals bioavailability; Flow Mediated Vasodilation; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active1 (Active Comparator): watermelon rind
  Interventions: Dietary Supplement: Watermelon Rind
- Active2 (Active Comparator): watermelon flesh
  Interventions: Dietary Supplement: Watermelon Flesh
- Active3 (Active Comparator): watermelon seeds
  Interventions: Dietary Supplement: Watermelon Seeds
- Control Comparator (Placebo Comparator): placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Watermelon Rind — watermelon rind
  Arms: Active1
Dietary Supplement: Watermelon Flesh — watermelon flesh
  Arms: Active2
Dietary Supplement: Watermelon Seeds — watermelon seeds
  Arms: Active3
Dietary Supplement: Placebo — Control Comparator
  Arms: Control Comparator

SUMMARY:
The primary objectives of the study are outlined below:

1. To investigate the relative bioavailability and absorption/kinetic profile of polyphenols after consumption of watermelon rind, flesh and seeds, respectively in an acute pilot study.
2. To study the effects of watermelon intake on endothelial function using the FMD technique and to understand the relationship between plasma metabolites, including L-citrulline and arginine, and FMD responses.

DETAILED DESCRIPTION:
The proposed trial will be a randomized, 4 arm, placebo controlled, within-subject crossover, study design. It is a pilot trial to establish methods and collect the preliminary data (N=6). Subjects meeting eligibility criteria (see eligibility criteria) will participate in 4 study visits where they will receive one serving (equivalent to 100 kcal) of 1 of 4 treatments: watermelon rind, watermelon flesh, watermelon seeds or placebo.

Qualified subjects from the screening visit will be randomized into the study and provided with a standard breakfast consisting of a high carbohydrate and moderate fat western-type meal 3 hours after the treatment. Each subject will be asked to come for one screening visit, a pre-study visit, and four dinner pick-ups on the day before each of the four test visits. The study day visit will last for approximately 9 h with a follow up visit the next day (24 h) for blood collection to allow for the characterization of target watermelon polyphenols and metabolites in plasma. Subjects will be instructed not to alter their usual diet or fluid intake during the study periods. Seven days prior to each study day visit, subjects will be advised not to consume fruits and vegetables rich in polyphenols and carotenoids or other high phytochemical foods (watermelon and products, arugula, spinach, tea, berries, grapes, carrots, tomatoes, sweet potatoes etc.).

Each study visit will involve with blood samples collection at time points 0 (fasting), 0.5, 1, 2, 3, 4, 5, 6, 7, 8 h and 24 hour (h). An assigned test treatment will be provided immediately after the 0 h blood collection, a breakfast meal will be provided immediately after the 2 h blood collection, and lunch after 6 h blood collection. FMD will be measured at 0 (fasting), 1, 3, 5, and 7h.

ELIGIBILITY:
Inclusion Criteria:

* • Men or women, 20-45 years of age with body mass index (BMI) in range from 27.5-32 kg/m2

  * Nonsmokers (Past smokers can be allowed if they have abstinence for minimum of 2 years)
  * No clinical evidence of cardiovascular, metabolic, respiratory, renal, gastrointestinal or hepatic disease
  * Not taking any medications that would interfere with outcomes of the study, i.e. lipid lowering medications, anti-inflammatory drugs, dietary supplements especially arginine and L-citrulline, etc.
  * Able to provide informed consent
  * Able to comply and perform the procedures requested by the protocol (including dietary restrictions, consumption of study treatments, records of food diary and questionnaire, and study visit schedule)

Exclusion Criteria:

* • Men and women who smoke

  * Men and women with known or suspected intolerance, allergies or hypersensitivity to study foods or treatments
  * Men and women who consume > 2 servings of watermelons per day
  * Men and women known to have/diagnosed with diabetes mellitus
  * Men and women who have fasting blood glucose concentrations > 125 mg/dL
  * Men and women who have uncontrolled blood pressure >140 mmHg (systolic)/90 mmHg (diastolic)
  * Men and women with documented vascular disease, e.g., heart failure, myocardial infarction, stroke, angina, related surgeries, etc. that, in the opinion of the investigator, could interfere with the interpretation of the study results
  * Men and women with cancer other than non-melanoma skin cancer in previous 5 years
  * Men and women diagnosed with chronic constipation, diarrhea or other chronic gastrointestinal complaint (e.g. irritable bowel syndrome)
  * Women who are known to be pregnant or who are intending to become pregnant over the course of the study
  * Women who are lactating
  * Taking medication or dietary supplements that may interfere with the outcomes of the study; e.g., antioxidant supplement, anti-inflammation, lipid lowering medication, blood pressure lowering medication, etc... Subjects may choose to go off dietary supplements (requires 30 days washout); e.g., fish oil, probiotics, etc...
  * Men and women who have donated blood within 3 months of the Screening Visit and blood donors/participants for whom participation in this study will result in having donated more than 1500 milliliters of blood in the previous 12 months.
  * Men and women who are vegans or vegetarian
  * History of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, or binge eating) diagnosed by a health professional
  * Substance (alcohol or drug) abuse within the last 2 years
  * Excessive coffee and tea consumers (> 5 cups/d)
  * Men and women who do excessive exercise regularly or an athlete
  * Unstable weight: gained or lost weight +/- 5 kg (11 lbs) in previous 2 months
  * Women who are taking unstable dose of hormonal contraceptives and/or stable dose for less than 6 months
  * Unusual working hours i.e., working overnight (e.g. 3rd shift)

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Quantitative characterization of watermelon polyphenolic compounds in plasma over 24-hour in humans | 24-hour Postprandial period
  This will be conducted by using ultra-high performance liquid chromatography iFunnel quadrupole time of flight mass spectrometer (UHPLC-QTOF-MS) and triple quadrupole mass spectrometer (UHPLC-QQQ-MS).

SECONDARY OUTCOMES:
The changes in endothelial function using ultrasound technique after consumption of each treatment | 24-hour Postprandial period
  Flow Mediated Vasodilation imaging of the brachial artery to assess endothelial-dependent relaxation
the relationship between plasma metabolites and FMD responses after consumption of treatments | 24-hour Postprandial period
  Correlation between plasma metabolites and FMD Change

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, Ph.D, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No